CLINICAL TRIAL: NCT03300674
Title: Intravenous Lidocaine Versus Hydromorphone for Acute Abdominal Pain. A Randomized Trial
Brief Title: Intravenous Lidocaine Randomized Comparative Effectiveness Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-8408
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Results first posted 2019-11-26 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain | interventions — Hydromorphone; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous hydromorphone (Active Comparator): Intravenous hydromorphone 1mg. A second dose can be administered at 30 minutes.
  Interventions: Drug: Hydromorphone
- Intravenous lidocaine (Active Comparator): Intravenous lidocaine 120 mg. A second dose can be administered at 30 minutes
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Hydromorphone — Hydromorphone intravenous infusion
  Arms: Intravenous hydromorphone
Drug: Lidocaine — Lidocaine intravenous infusion
  Arms: Intravenous lidocaine

SUMMARY:
This is a randomized, double-blind, emergency department based, comparative effectiveness study of two medication for acute abdominal pain: intravenous lidocaine and intravenous hydromorphone. Patients will be enrolled during an emergency department visit and followed throughout their emergency department course and then by telephone 7 days later.

ELIGIBILITY:
Inclusion Criteria:Eligible patients are those who present to an ED for treatment of acute abdominal pain. Acute will be defined as pain for no more than seven days. At the time of enrollment, the ED treatment plan must include use of an intravenous opioid.

Exclusion Criteria: Patients will be excluded from participation if they have cardiac conduction system impairment (QTc duration > 0.5s, QRS duration > 0.12s, or PR interval duration > 0.2s), known renal (CKD >2) or liver disease (Childs-Pugh B or greater), are hemodynamically unstable, as determined by the attending physician, are pregnant or breastfeeding, or have a known allergy to either medication. Patients will also be excluded if they have used prescription or illicit opioids within the previous week, or if they have a chronic pain disorder, defined as use of any analgesic medication on more days than not during the month preceding the acute episode of pain. Patients weighing < 60kg or > 120kg will be excluded.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chinn E, Friedman BW, Naeem F, Irizarry E, Afrifa F, Zias E, Jones MP, Pearlman S, Chertoff A, Wollowitz A, Gallagher EJ. Randomized Trial of Intravenous Lidocaine Versus Hydromorphone for Acute Abdominal Pain in the Emergency Department. Ann Emerg Med. 2019 Aug;74(2):233-240. doi: 10.1016/j.annemergmed.2019.01.021. Epub 2019 Feb 26. PMID 30819520

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Hydromorphone | Intravenous Lidocaine
Started | 77 | 77
Completed | 77 | 77
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Hydromorphone | Intravenous Lidocaine | Total
Number analyzed (Participants) | 77 | 77 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (13) | 42 (12) | 41 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 54 | 98
  Male | 33 | 23 | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 77 | 77 | 154
Pain duration in days [Median (Inter-Quartile Range); unit: days] | 2 [1 to 3] | 2 [1 to 4] | 2 [1 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Change in 0-10 Pain Scale Between Baseline and 90 Minutes
Description: Participants were asked to describe their pain on a scale from 0 to 10 with 0= no pain and 10= the worst pain imaginable
Time Frame: up to 90 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Hydromorphone | Intravenous Lidocaine
Number analyzed (Participants) | 77 | 77
units on a scale | 5.0 (2.8) | 3.8 (2.2)

2. Secondary Outcome: Rescue Medication
Description: no need for off-protocol parenteral pain medication during the ED visit. The following parenteral medications will be considered off protocol pain medication: any opioid, any non-steroidal anti-inflammatory drug
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Hydromorphone | Intravenous Lidocaine
Number analyzed (Participants) | 77 | 77
Participants | 20 | 39

3. Secondary Outcome: Adverse Events
Description: Any new symptom development after administration of investigational medication
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Hydromorphone | Intravenous Lidocaine
Number analyzed (Participants) | 77 | 77
Participants | 28 | 23

ADVERSE EVENTS:
Time Frame: 3 hours
Arm/Group | Intravenous Hydromorphone | Intravenous Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/77
Other Adverse Events (participants affected / at risk) | 28/77 | 23/77
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Hydromorphone (N=77) | Intravenous Lidocaine (N=77)
dizziness (Nervous system disorders) | 14 (14) | 4 (4)
drowsiness (Nervous system disorders) | 6 (6) | 4 (4)
headache (Nervous system disorders) | 3 (3) | 6 (6)
nausea (Gastrointestinal disorders) | 13 (13) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT03300674/Prot_SAP_001.pdf